CLINICAL TRIAL: NCT03611348
Title: Effectiveness of Microneedling and Topical Latanoprost in Treatment of Acrofacial Vitiligo
Brief Title: Microneedling and Latanoprost in Acrofacial Vitiligo
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Noreen Ismail AbdelGhani Ahmed, resident at general administration of medical affairs, Sohag University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIT.LT2018
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Vitiligo
Keywords: acrofacal vitiligo, latanoprost, microneedling
MeSH Terms: conditions — Vitiligo | interventions — Latanoprost; Percutaneous Collagen Induction

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Microneedling + latanoprost (Active Comparator): patient will receive topical application of latanoprost 0.005% eye drops solution twice daily for 3 months preceded by microneeding in sessions by dermapen every 2 weeks for 3 months (totally 6 sessions).
  Interventions: Drug: Latanoprost; Device: Microneedling
- latanoprost (Active Comparator): Patient will receive topical application of latanoprost 0.005% eye drops solution only twice daily for 3 months (active control side).
  Interventions: Drug: Latanoprost

INTERVENTIONS:
Drug: Latanoprost — Topical application of latanoprost 0.005% eye drops solution only twice daily for 3 months.
  * To apply latanoprost solution, one drop of the solution will be distributed over 1cm2 of depigmented skin. Side effects will be recorded.
Device: Microneedling — A superficial micro-needling technique will be done in millimeters according to depth of skin. The vitiliginous area and a thin surrounding rim (about 2 mm) will be subjected to micro-needling with dermapen. The depth of abrasion will be guided by the depth adjustor according to depth of skin on the affected area. This will be followed by the appearance of multiple, tiny, punctate, bleeding points
  Arms: Microneedling + latanoprost

SUMMARY:
To compare efficacy of topical latanoprost preceded by microneedling versus topical latanoprost alone in treatment of acrofacial vitiligo.

DETAILED DESCRIPTION:
patients meeting inclusion and exclusion criteria presented to Dermatology Outpatient Clinic, Sohag University Hospital will be enrolled in the study after obtaining a written consent from them. Full history will be obtained and meticulous examination will be carried out. Patients will be randomly divided into 2 groups, one group will receive topical latanoprost with microneedling, and the other one will receive topical latabnoprost alone.

ELIGIBILITY:
Inclusion Criteria:

- Acrofacial stable vitiligo for 6 months duration (without new lesions appearance or change in size of the existing lesions).

Exclusion Criteria:

* History of scar formation.
* Patients with systemic diseases (diabetes, bleeding disorders, chronic renal diseases, chronic liver diseases, asthma and hypertension).
* Patients who are receiving chemotherapy or radiotherapy.
* Pregnant and lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in VASI score | 6 months
  VASI score: The percentage of vitiligo involvement is calculated in terms of hand units. One hand unit is approximately equivalent to 1% of the total body surface area. The degree of pigmentation is estimated to the nearest of one of the following percentages:
  * 100% - complete depigmentation, no pigment is present
  * 90% - specks of pigment present
  * 75% - depigmented area exceeds the pigmented area
  * 50% - pigmented and depigmented areas are equal
  * 25% - pigmented area exceeds depigmented area
  * 10% - only specks of depigmentation present. The VASI for each body region is determined by the product of the area of vitiligo in hand units and the extent of depigmentation within each hand unit measured patch.
  Total body VASI = S All body sites [Hand Units] x [Residual depigmentation]. (Feily et al., 2014).

CONTACTS AND LOCATIONS:
Overall Officials: Ramadan Saleh, MD, Study Director — Sohag University

IPD SHARING:
Plan to Share IPD: Yes
Share study proposal, patients and methods, results.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 1 year
Access Criteria: Permission obtained from study director